CLINICAL TRIAL: NCT03798314
Title: Phase I Clinical Trial for Evaluation of Nivolumab and Pomalidomide Combination for Relapsed/Refractory Primary Central Nervous System Lymphoma and Primary Vitreoretinal Lymphoma
Brief Title: Nivolumab and Pomalidomide in Treating Patients With Relapsed or Refractory Central Nervous System Diffuse Large B Cell Lymphoma or Primary Vitreoretinal Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC178A; NCI-2018-03661 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC178A (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2019-01-02; First posted 2019-01-09 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Nervous System Lymphoma; Recurrent Primary Vitreoretinal DLBCL; Refractory Nervous System Lymphoma; Refractory Primary Vitreoretinal DLBCL
MeSH Terms: interventions — Nivolumab; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nivolumab and pomalidomide) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and pomalidomide PO on days 1-14. Treatment repeats every 4 weeks until disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Pomalidomide

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase I trials studies side effects and best dose of pomalidomide when given together with nivolumab in treating patients with primary central nervous system diffuse large B cell lymphoma or primary vitreoretinal diffuse large B cell lymphoma that has come back or that has not responded to treatment. Immunotherapy with monoclonal antibodies, such as pomalidomide and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of pomalidomide which can be safely combined with the fixed dose schedule of nivolumab in patients with relapsed/refractory primary central nervous system lymphoma (PCNSL) and primary vitreoretinal lymphoma (PVRL). (Phase I)

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) and progression free survival (PFS) of nivolumab and pomalidomide combination in patients with relapsed/refractory PCNSL and PVRL.

OUTLINE: This is dose-escalation study of pomalidomide.

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and pomalidomide orally (PO) on days 1-14. Treatment repeats every 4 weeks until disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 weeks, then every 3 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have one of the following:

  * Relapsed or refractory primary central nervous system (CNS) diffuse large B cell lymphoma (PCNSDLBCL) with a brain lesion >= 1 cm, or with cerebrospinal fluid (CSF) relapse with positive CSF cytology, or with ocular relapse with positive ocular tissue biopsy

    * NOTE: Tissue biopsy is not absolutely necessary for brain tumor unless clinical and radiologic findings strongly suggest other etiologies as per treating physician. Initial diagnosis must be made by tissue biopsy OR
  * Relapsed/refractory primary vitreoretinal diffuse large B cell lymphoma (DLBCL) with a CNS lesion >= 1 cm, or with CSF relapse with positive CSF cytology, or with ocular relapse with positive ocular tissue biopsy. Relapsed PVRL must have progressed or failed at least one systemic regimen

    * NOTE: Intraocular treatments are not regarded as systemic therapy
    * NOTE: If recurrence in ocular or leptomeningeal space, the patient will need a positive ocular tissue biopsy and CSF biopsy. Tissue biopsy requirement of the CNS lesion is as outlined in bullet above
* Patient progressed after or did not respond to at least 1 line of systemic therapy (e.g., high-dose methotrexate, high-dose methotrexate based regimen, high dose cytarabine, etc)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2 or 3
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 (within =< 14 days prior to registration)
* Hemoglobin >= 9.0 g/dL (within =< 14 days prior to registration)
* Direct bilirubin < 1.5 x upper limit of normal (ULN) (or total bilirubin =< 3.0 x ULN with direct bilirubin =< 1.5 x ULN in patients with well-documented Gilbert?s Syndrome) (within =< 14 days prior to registration)
* Aspartate transaminase (AST) =< 3 x ULN (within =< 14 days prior to registration)
* Creatinine =< 1.5 x ULN OR calculated creatinine clearance must be >= 45 ml/min using the Cockcroft-Gault formula (within =< 14 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of anticoagulants (within =< 14 days prior to registration)
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/ml, =< 14 days prior to registration and within 24 hours of starting pomalidomide. In addition, must either commit to continue abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. WOCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a WOCBP even if they have had a vasectomy. In addition, women of childbearing potential (WOCBP) receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of nivolumab. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure

  * A woman of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Able to take aspirin (81 or 325 mg) daily or an anticoagulant (as determined by treating physician) as prophylactic anticoagulation
* Provide written informed consent
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to undergo biopsy procedures, if deemed necessary by treating physician
* Willing to be registered into a mandatory POMALYST REMS program, and willing and able to comply with the requirements of the POMALYST REMS program

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Other active malignancy =< 3 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not have received immune checkpoint inhibitors or immunomodulatory therapy (IMiD) for their cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Use of corticosteroid in the absence of cerebral edema

  * NOTE: If a corticosteroid is used, it should be used at the lowest dose possible for the shortest possible duration. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of treatment assignment are excluded
  * EXCEPTIONS: Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Therapy with myelosuppressive chemotherapy or biologic therapy =< 21 days prior to registration with incomplete recovery of blood counts
* Persistent toxicities >= grade 3 from prior chemotherapy or biological therapy regardless of interval since last treatment
* History of thromboembolic episodes =< 3 months prior to registration
* Active hepatitis B or C with uncontrolled disease

  * NOTE: A detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients. Hepatitis B core IgM antibody (HBcIgM Ab), Hepatitis B surface antigen (HBsAg) and Hepatitis C virus (HCV) Ab screen (Scrn) w/Reflex testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV infection
* Inability to swallow or impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) that would preclude use of oral medications
* Major surgery =< 4 weeks prior to registration or have not recovered from side effects of such therapy
* New York Heart Association classification III or IV
* Patient received radiation alone previously

  * NOTE: Radiation therapy would not be regarded as a systemic therapy
  * EXCEPTION: Patients who have received systemic therapy followed by radiation would be eligible
* PCNSL with systemic disease
* Inability to undergo or have a magnetic resonance imaging (MRI) performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of pomalidomide | Up to 28 days
  The MTD in this study will be defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients).
Incidence of adverse events | Up to 12 weeks following end of treatment.
  Will be evaluated by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number and severity of all adverse events will be tabulated and summarized in this patient population both overall and by dose level. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Percentage of Participants With Grade 3 or Higher Adverse Events Considered At Least Possibly Related to Treatment | Up to 12 weeks following end of treatment
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 4 years
  Will be estimated by the number of patients with an objective status of complete response (CR), unconfirmed complete response (CRu), or partial response (PR) divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Progression-free survival (PFS) | From registration to progression or death due to primary central nervous system lymphoma (PCNSL) or primary vitreoretinal lymphoma (PVRL), assessed up to 4 years
  Will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 12 weeks following treatment
  Will be assessed by CTCAE version 5.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Han Tun, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota